CLINICAL TRIAL: NCT03535636
Title: Sleep Impairments in Refugees Diagnosed With PTSD - A Polysomnographic and Self-report Study
Brief Title: Sleep Impairments in Refugees Diagnosed With PTSD
Acronym: PSG-PTSD
Status: Completed | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Danish Center for Sleep Medicine (Other)
Responsible Party: Principal Investigator, Mia Beicher Ansbjerg, Pregraduate Researcher, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Other Study IDs: PSG-PTSD
Record Dates: First submitted 2018-04-24; First posted 2018-05-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: PTSD; Sleep Disorder
Keywords: Polysomnography; Refugees
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Refugees with PTSD: Adults over the age of 18. Refugees or family members of refugees that has been reunited. PTSD (ICD-10 criteria) and written consent.
  No drug or alcohol abuse and no medication that can affect sleep rhythms, such as antipsychotic drugs, benzodiazepine, opioids, antihistamine or CNS stimulating drugs.
  A BMI under 35 and no pregnancy.
  Interventions: Other: Polysomnography
- Healthy controls: Matched on age, sex and BMI and signed written consent. No mental illness, drug or alcohol abuse and medication. No pregnancy.
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — Sleep architecture will be assessed by polysomnography

SUMMARY:
The aim of this study is to examine sleep architecture in refugees with PTSD. Polysomnography (PSG) will be carried out to study the occurrence of sleep disorders in patients and healthy controls.

DETAILED DESCRIPTION:
There is little knowledge on treatment of sleep disturbances in trauma-affected refugees and this study will be the first to record the biophysiological changes that occur during sleep in refugees with PTSD. The study is a proof-of-concept study and this will contribute with new and potentially crucial knowledge of sleep disturbances in these patients.

The project is designed as a cross-sectional study with 20 refugees with PTSD referred to the specialised outpatient clinic, Competence Centre for Transcultural Psychiatry (CTP), and 20 healthy control subjects.

All patients referred to CTP will be invited to an initial consultation with a doctor. During this consultation a diagnostic assessment will be performed and the clinical history will be obtained. Patients who give informed consent will be invited to participate in the project and have sleep measurements performed by PSG. Furthermore self-administered questionnaires and semi-structured interviews will be used to collect information on mental health, sleep quality, sleep length and nightmares.

Each patient will be equipped with PSG equipment to do measurements at home for one night (12 hours). Healthy control subjects will fill out the same CTP standard ratings and have the same diagnostic assessment and PSG measurement.

The hypothesis is that the sleep architecture in refugees with PTSD differ from healthy controls. It is suggested that refugees with PTSD have increased dream activity as well as increased incidence of sleep disorders such as rapid eye movement (REM) sleep without atonia (RSWA), REM sleep behaviour disorder (RBD), sleep apnea and periodic limb movement disorder (PLM).

The study is performed in collaboration with Danish Centre for Sleep Medicine in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years old or above)
* Refugee or family reunification refugees
* PTSD according to the ICD-10 criteria's
* Signed informed concent

Exclusion Criteria:

* Severe psychotic disorder (defined as patients with ICD-10 diagnoses F2x and F30.1-F30.9)
* Harmful use of alcohol (ICD-10 diagnosis F1x.1)
* Serious or progressive somatic illnesses that the lead investigator finds interfering for the study
* Medical treatment with antipsychotics, benzodiazepine, opioids, CNS stimulants or regular use of anti histamine
* BMI >35
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes patients referred to the specialised outpatient clinic 'Competence Centre for Transcultural Psychiatry' (CTP) in Denmark. The clinic treats adult refugees, migrants or people with family reunification who has a traumatic background eg. imprisonment with torture, organised violence, long term political pursuit or war experiences. The patients at the clinic has PTSD, depression and/or anxiety.
  Healthy control subjects are matched on age, sex and BMI.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Assessing the incidence of sleep disorders in refugees with PTSD | 12 hours
  Sleep architecture will be assessed by polysomnography. The recording of brain activity during sleep will reveal the incidence of sleep disorders such as sleep apnea, REM sleep without atonia and REM sleep behaviour disorder

SECONDARY OUTCOMES:
Global Assessment of Functioning (GAF S + F) | 10 minutes
  A numeric scale used to subjectively rate the social, occupational, and psychological functioning of an individual
Harvard Trauma Questionnaire (HTQ) | 10 minutes
  Assessing PTSD symptoms
Hopkins Symptom Check List-25 (HSCL-25) | 10 minutes
  Assessing anxiety and depression symptoms
World Health Organization Well-Being Index (WHO-5) | 10 minutes
  Assessing subjective psychological well-being
Sheehan Disability Scale (SDS) | 10 minutes
  The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. Total score 0-30 (0 unimpaired, 30 highly impaired). Work/school (0-10), Social life (0-10), Family life/home responsibilities (0-10). Scores of ≥5 on any of the 3 scales; high scores are associated with significant functional impairment.
Schedule for Clinical Assessment in Neuropsychiatry (SCAN) | 1 hours
  Diagnosing and measuring mental illness that may occur in adult life.
Clinician Administered PTSD Scale (CAPS-5) | 1 hour
  Assessing PTSD symptoms, including their frequency and severity. The gold standard in PTSD assessment. The CAPS-5 is a 30-item structured interview and requires the identification of a single index trauma to serve as the basis of symptom inquiry. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. Similarly, CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). A symptom cluster score may also be calculated for dissociation by summing items 19 and 20. A patient needs to have: at least one Criterion B and C symptom and at least two Criterion D and E symptoms. Criterion F is met (disturbance has lasted one month) and Criterion G is met (disturbance causes either clinically significant distress or functional impairment).
Hamilton depression scale (HAM-D17) | 15 minutes
  Assessing a patient's severity of depression before, during, and after treatment. The HAM-D probes 17 parameters. Some items are scored on a 5-point scale, ranging from 0=not present to 4=severe; others are scored on a 3-point scale, ranging from 0=not present to 2=severe. Total score 0-52 (0 unimpaired, 52 highly impaired). The sum of all 17 items indicate the severity of depression; 0-12 = normal, 13-17 = mild depression, 18-24 = moderate depression, 24-52 severe depression.
Hamilton anxiety scale (HAM-A14) | 15 minutes
  Assessing the severity of a patient's anxiety. The HAM-A probes 14 items. Each item is scored on a 5-point scale, ranging from 0=not present to 4=severe. Total score 0-56 (0 unimpaired, 56 highly impaired). The sum of all 14 items indicate the severity of anxiety; 14-17 = mild anxiety, 18-24 = moderate anxiety, 25-30 severe anxiety.
The Pittsburgh Sleep Quality Index (PSQI) | 10 minutes
  Assessing sleep quality and sleep disorders
Disturbing dreams and Nightmare Severity Index (DDNSI) | 10 minutes
  Assessing nightmares
REM Sleep Behavior Disorder Screening Questionnaire (RBDSC) | 10 minutes
  Assessing REM Sleep Behavior Disorders
Life Events Checklist for DSM-5 (LEC-5) - extended version | 10 minutes
  Screening of potential traumatic events

CONTACTS AND LOCATIONS:
Locations (1):
- Competence Center for Transcultural Psychiatry, Ballerup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ansbjerg MB, Sandahl H, Baandrup L, Jennum P, Carlsson J. Sleep impairments in refugees diagnosed with post-traumatic stress disorder: a polysomnographic and self-report study. Eur J Psychotraumatol. 2023;14(1):2185943. doi: 10.1080/20008066.2023.2185943. PMID 36971225